CLINICAL TRIAL: NCT05450380
Title: Clinical Investigation to Assess Safety and Performance of Dermal Filler of Hyaluronic Acid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mesoestetic Pharma Group S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-LIFT001-042022
Record Dates: First submitted 2022-06-15; First posted 2022-07-08 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Skin Folds; Wrinkle

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: LIFT001 (Experimental): LIFT001 is composed by sodium hyaluronate at concentration of 2,5% (25 mg/ml) with 1,4-Butanediol diglycidyl ether (BDDE) acting as a cross-linking agent, in aqueous solution at physiological pH. The filler of 1ml is administered once or twice depending on the individual necessity.
  The dermal filler of hyaluronic acid LIFT001 is applied to the facial area to provide firmness and counteract sagging for the correction of deep wrinkles and imperfections of face.
  Interventions: Device: LIFT001

INTERVENTIONS:
Device: LIFT001 — The dermal filler of hyaluronic acid LIFT001 is applied to the facial area to provide firmness and counteract sagging for the correction of deep wrinkles and imperfections of face.
  The dermal filler of hyaluronic acid LIFT001 is applied to the facial area to provide firmness and counteract sagging for the correction of deep wrinkles and imperfections of face.

SUMMARY:
The objective of this clinical investigation is to assess the safety and performance of dermal filler of hyaluronic acid to provide firmness and counteract sagging for the correction of deep wrinkles and imperfections in the lower two thirds of the face at 2 months post-treatment.

DETAILED DESCRIPTION:
The primary endpoint is to assess the safety of dermal filler of hyaluronic acid by occurrence of Treatment-Related Adverse Events (TRAEs) and Serious Adverse Events (SAEs) through 2 months post-treatment. Furthermore, the performance of the device will also be assessed as the aesthetical outcome measured by the Global Aesthetic Improvement Scale (GAIS), Wrinkle Severity Rating Scale (WSRS), and 2D images of subjects' faces at 2 months post-treatment.The secondary endpoints are the following:

Secondary Safety Endpoint

* To assess the safety of dermal filler of hyaluronic acid by occurrence of Treatment-related Adverse Events (TRAEs) and Serious Adverse Events (SAEs) through 6-, 9-, and 12-months post-treatment.
* To assess the safety of dermal filler of hyaluronic acid by occurrence of all AEs through 2-, 6-, 9-, and 12-months post-treatment.

Secondary Performance Endpoint

* To evaluate the performance of dermal filler of hyaluronic acid at 6-, 9- and 12-months post-treatment, assessed as the aesthetical outcome measured by the Global Aesthetic Improvement Scale (GAIS)
* Assessment of dermal filler of hyaluronic acid performance of mesofiller® Lift at 6-, 9- and 12-months post-treatment using the Wrinkle Severity Rating Scale (WSRS)
* Assessment of dermal filler of hyaluronic acid performance of dermal filler of hyaluronic acid at 6-, 9- and 12-months post-treatment using 2D images of subjects' faces
* Assessment of dermal filler of hyaluronic acid performance of dermal filler of hyaluronic acidt at 6-, 9- and 12-months post-treatment through satisfaction surveys related to the subject's appearance.

ELIGIBILITY:
Inclusion Criteria:

1. Subject who had provided written informed consent form.
2. Adult male or female subjects between 45 and 70 years old.
3. Subject with moderate (2) or higher score in the Wrinkle Severity Rating Scale (WSRS) in the lower two thirds, and in at least one of the two sides of the face, assessed at baseline by the treating investigator.
4. Subject must be willing to abstain from any other facial invasive treatment (plastic surgery, implants, peelings) in the lower two thirds of the face during the clinical investigation period.

Exclusion Criteria:

1. History of severe or multiple allergies, including allergy or hypersensitivity to injectable hyaluronic acid gel, lidocaine, anesthetics, or nerve-blocking agents or any of the components of product.
2. Any disease at baseline that results in changes of facial contour or facial edema.
3. Active skin disease or inflammation on or near the injection area at baseline that could interfere with the clinical investigation injections or assessments.
4. History of connective tissue diseases.
5. Soft tissue augmentation in the previous 6 months with bovine collagen, in the previous 12 months with porcine or human collagen, or in the previous 18 months with hyaluronic acid or hydroxyapatite.
6. Any aesthetic treatment/procedure on the face in the previous 6 months that may interfere with study injections and/or study assessments.
7. Subjects who have received permanent facial implants within the previous 36 months.
8. Presence of any condition, which in the opinion of the investigator, made the subject unable to complete the clinical investigation per protocol.
9. Subjects who are currently participating in another clinical investigation which may interfere with this clinical investigation.
10. Pregnant or nursing subjects, and subjects who plan pregnancy during the clinical investigation period.
11. Subjects undergoing restrictive nutritional regimens.
12. Subjects who practice facial impact sports, such as boxing, karate, taekwondo and other similar sports.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of occurrence of Treatment-Related Adverse Events (TRAEs) and Serious Adverse Events (SAEs) of device LIFT001 at 2 months time | 2 MONTHS
  The primary endpoint is to assess the safety of product LIFT001 by occurrence of Treatment-Related Adverse Events (TRAEs) and Serious Adverse Events (SAEs) through 2 months post-treatment.
Performance of device LIFT001 at 2 months time - GAIS scale | 2 MONTHS
  The performance of the device LIFT001 will also be assessed as the aesthetical outcome measured by:
  * Global Aesthetic Improvement Scale (GAIS)
  Score Grade Description 7 Very Much Improved Very marked improvement in appearance to
  1 Very Much Worse The appearance is very much worse than the original condition
Performance of device LIFT001 at 2 months time - WSRS scale | 2 MONTHS
  The performance of the device LIFT001 will also be assessed as the aesthetical outcome measured by:
  - Wrinkle Severity Rating Scale (WSRS)
  Score Severity descriptions 4 Extreme Very deep wrinkle, redundant fold (overlapping skin) 0 None No wrinkle
Performance of device LIFT001 at 2 months time - 2D images | 2 MONTHS
  The performance of the device LIFT001 will also be assessed as the aesthetical outcome measured by:
  - 2D images of subjects' faces at 2 months post-treatment.

SECONDARY OUTCOMES:
Evaluation of occurrence of Treatment-Related Adverse Events (TRAEs) and Serious Adverse Events (SAEs) of device LIFT001 at 6, 9 and 12 months time | 12 MONTHS
  * To assess the safety of LIFT001 by occurrence of Treatment-related Adverse Events (TRAEs) and Serious Adverse Events (SAEs) through 6-, 9-, and 12-months post-treatment.
  * To assess the safety of LIFT001 by occurrence of all AEs through 2- , 6-, 9-, and 12-months post-treatment.
Performance of device LIFT001 at 12 months time - GAIS scale | 12 months
  To evaluate the performance of LIFT001 at 6-, 9- and 12-months post-treatment, assessed as the aesthetical outcome measured by:
  - Global Aesthetic Improvement Scale (GAIS) Score Grade Description 7 Very Much Improved Very marked improvement in appearance to
  1 Very Much Worse The appearance is very much worse than the original condition
Performance of device LIFT001 at 12 months time - WSRS scale | 12 months
  To evaluate the performance of LIFT001 at 6-, 9- and 12-months post-treatment, assessed as the aesthetical outcome measured by:
  - Wrinkle Severity Rating Scale (WSRS) Score Severity descriptions 4 Extreme Very deep wrinkle, redundant fold (overlapping skin) 0 None No wrinkle
Performance of device LIFT001 at 12 months time - 2D images | 12 months
  To evaluate the performance of LIFT001 at 6-, 9- and 12-months post-treatment, assessed as the aesthetical outcome measured by:
  - 2D images of subjects' faces at 6, 9 and 12 months post-treatment.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Centro Dermatologico Internacional - Cdi, Madrid, CAM
  - Hospital Ruber Internacional, Madrid, CAM